CLINICAL TRIAL: NCT04376190
Title: Three-dimensional Judgment of Mandibular Condylar Volume and Position Subsequent to Twin-block Functional Therapy of Skeletal Class II Malocclusion Accompanied With Low-level Laser Therapy
Brief Title: Effect of Low Level Laser Therapy on the Temporomandibular Joint During Treatment of Skeletal Class II Malocclusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mahmoud abdelhameed mohamed (Other)
Responsible Party: Sponsor-Investigator, mahmoud abdelhameed mohamed, Dentist, Ministry of Health, Egypt, MSc studentDepartment of Orthodontics, Faculty of Dental Medicine (Boys), Al-Azhar University, Cairo, Egypt., Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlAzharU 7712
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Malocclusion Class II
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: laser group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): 12 patients treated with twin block functional appliance without low-level laser application for 9 month
- laser group (Experimental): 12 patients treated with twin block functional appliance with low-level laser application with the following set parameters; 635 nm wavelength in continuous-wave mode, 50 mw power output, 4.5 J/cm2 energy density, 11.25 J total dose per side, 45 seconds/ point, and 8 mm fiber optic tip diameter. The laser was applied at five points located within TMJ region on both right and left sides in contact with skin as follows: lateral, superior, anterior, posterior, and posterior- inferior points. Laser application was repeated weekly for three months according to a standard protocol
  Interventions: Radiation: low level laser therapy

INTERVENTIONS:
Radiation: low level laser therapy — In the laser group, patients received LLLT from a semiconductor Gallium Aluminum Arsenide diode laser (SMARTMPRO, LASOTRONIX, Poland) with the following set parameters; 635 nm wavelength in continuous-wave mode, 50 mw power output, 4.5 J/cm2 energy density, 11.25 J total dose per side, 45 seconds/ point, and 8 mm fiber optic tip diameter. Laser was applied (Fig.2) at five points located within TMJ region on both right and left sides in contact with skin as follows: lateral, superior, anterior, posterior, and posterior- inferior points.
  Other Names: photobiomodulation
  Arms: laser group

SUMMARY:
to evaluate effect of low-level laser therapy (LLLT) on mandibular condylar volume and position after treatment of Class II malocclusion with Twin Block (TB) functional therapy via cone beam computed tomography (CBCT).

Materials and methods: Twenty eight growing patients, 14 boys and 14 girls ranged in age 9-12 years, were randomly divided into control group (mean initial age 10.64±1.36 years) and laser group (mean initial age 10.55 1.45 years). All patients treated with TB appliance where Gallium aluminum arsenide diode laser applied in one group weekly around TMJ region for 12 sessions in three months with set parameters: continuous 635 nm, 50 mW, 4.5J/cm2, 45 seconds/ point, total dose per side 11.25J. CBCT were obtained before and immediately after TB therapy, in addition to routine orthodontic records. Changes in TMJ and skeletal variables were analyzed and compared within and between both groups.

DETAILED DESCRIPTION:
to evaluate the effect of low-level laser therapy (LLLT) on mandibular condylar volume and position after treatment of Class II malocclusion with Twin Block (TB) functional therapy via cone-beam computed tomography (CBCT).

Materials and methods: Twenty-eight growing patients, 14 boys, and 14 girls ranged in age 9-12 years, were randomly divided into control group (mean initial age 10.64±1.36 years), and laser group (mean initial age 10.55 1.45 years). All patients treated with TB appliance where Gallium aluminum arsenide diode laser applied in one group weekly around TMJ region for 12 sessions in three months with set parameters: continuous 635 nm, 50 mW, 4.5J/cm2, 45 seconds/ point, total dose per side 11.25J. CBCT were obtained before and immediately after TB therapy, in addition to routine orthodontic records. Changes in TMJ and skeletal variables were analyzed and compared within and between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Class II (ANB°> 5°) with the normal maxilla (SNA°=82°±4°) and retrognathic mandible (SNB°< 78°).
* Overjet greater than 5 mm.
* Minimal crowding in dental arches (≤ 3 mm).
* The lower incisors should be on average inclination or slightly retroclined.
* All the patients were in stages II and III based on the modified cervical vertebral maturation stages(CVMS) according to Bacetti et al.

Exclusion Criteria:

* Previous history of orthodontic treatment.
* Congenitally missing or extracted permanent tooth (except third molars).
* Posterior crossbites or severe maxillary transverse deficiency.
* Severe facial asymmetry determined by clinical or radiographic examination.
* Poor oral hygiene.
* Systemic diseases that may affect orthodontic treatment results.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Changes of condylar volume (mm3) and condylar head position before and after Twin-block therapy with and without LLLT: | after 9 mouth from starting treatment
  3D condylar volume measured using software and 2D condylar head position

SECONDARY OUTCOMES:
Changes of cephalometric skeletal measurements before and after Twin-block therapy with and without LLLT | after 9 mouth from starting treatment
  measured ANB, SNA, SNB effective mandibular, ramus, and corpus lengths

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A Mohamed, MSc student, Principal Investigator — Al-Azhar University
Locations (1):
- Faculty of Dental Medicine (Boys), Al- Azhar University,, Cairo, Cairo Nasr City, Egypt